CLINICAL TRIAL: NCT05021497
Title: Effects Of Global Postural Re-Education (GPR) On Patients With Non-Specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00941 Faisal Saeed
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Neck Pain
Keywords: Pain; Range of motion; Kinesiophobia; Forward head posture
MeSH Terms: conditions — Neck Pain; Pain; Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Positional Re-education (Experimental): Global Positional Re-education
  Interventions: Other: Global Positional Re-education
- Conventional Physical Therapy Program (Active Comparator): Conventional therapy will consist of a combination of manual techniques
  Interventions: Other: Conventional Physical Therapy Program

INTERVENTIONS:
Other: Global Positional Re-education — A series of gentle active movements and postures aimed at realigning joints and stretching shortened muscles. GPR includes 8 therapeutic postures in lying, sitting and standing.
  Arms: Global Positional Re-education
Other: Conventional Physical Therapy Program — Axial traction will be given for 5 minutes, followed by mobilization of the muscle fascia along with static stretching of the scalene, levator scapulae, upper trapezius, sternocleidomastoid and pectoralis minor muscles.
  Arms: Conventional Physical Therapy Program

SUMMARY:
Pain is an "unpleasant sensory and emotional experience (associated with actual or potential tissue damage". Chronic pain is a sensation of hyperalgia to muscles, ligaments and skin on both active and passive movements. Chronic pain has a tendency to prevent people from working and exercising

DETAILED DESCRIPTION:
Neck pain is a very common clinical condition which equals the economic, social cost and level of disability to that of low back pain.Mechanical neck pain that occurs without an identifiable underlying disease and anatomical abnormality is termed as "non-specific" neck pain (NS-NP).Mechanical neck pain commonly arises insidiously and is generally multifactorial in origin.Two most common complains associated with chronic specific and non-specific neck pain are Kinesiophobia (fear of movement) and Postural asymmetry (forward head posture). Medical, surgical and physical therapy treatments are recommended for addressing chronic non-specific neck pain. Within the scope of physical therapy conventional management consist of many different techniques such as therapeutic exercises, electrotherapy, Pilates, yoga and manual therapy. Manual therapy is among the most common used method for treating musculoskeletal conditions including chronic neck pain. Manual therapy consists of stretching techniques, joint mobilization/manipulation, isometric/dynamic strengthening exercises and fascial manipulation or release. Global Postural Re-education (GPR) is an alternative therapeutic strategy based on the concept that postural muscles are organized in the form of 'muscle chains' located on the anterior and posterior aspect of the spine. It involves the global stretching of the anti-gravitational muscles and the kinetic muscle chains.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific neck pain ≥ 3 months.
* No prior medication and Physical Therapy interventions from last 3 months.
* Pain: moderate level (6 on NPRS).

Exclusion Criteria:

* History of any trauma .
* History of any psychological condition.
* Specific causes of Neck Pain (e.g., systemic, rheumatic, neuromuscular diseases).
* Presence of central and peripheral neurological sign.
* Spinal surgery

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | six weeks
  The NPRS is an 11-point numeric scale, it is the segmented numeric version of the visual analog scale. Subjects will be asked to mark/select a whole number for 0-10 that best describes their perceived pain intensity of the last 24 hours. Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week
Neck Disability Index | six weeks
  it is a 10-item self-report questionnaire that measures the patient's disability related to his/her neck pain. It is the most commonly used questionnaire for neck disability; its reliability and validity has been demonstrated in many literatures and languages. Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week
Goniometer for Cervical Range of Motion | six weeks
  The active cervical range of motion (CROM) will be measured in sitting posture by using a universal goniometer, which consists of two arms; one that is stationary and one that is moveable. Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week
Tampa Scale of Kinesiophobia | six weeks
  Tampa Scale of Kinesiophobia (TSK). TSK is a 17-items questionnaire based on the evaluation of fear of movement, fear of physical activity and fear of re-injury in patients suffering from chronic musculoskeletal pain. It is the most widely used fear avoidance behavior questionnaire with good level of reliability and validity as documented in different literatures. TSK is composed of 17 items with score ranging from 1to 4 for each item, ultimately having a total score ranging from 17-68.Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week

SECONDARY OUTCOMES:
Forward Head Posture: | six weeks
  Ruler method. This method involves measuring the distance from the wall to the tragus of the ear (Tragus to wall test) and from wall to the posterior aspect of acromion of shoulder by a ruler in standing position. The normal distance of Tragus to wall (TTW) in males is 10.55 cm and in females is 10.00 cm, whereas the normal distance of shoulder from wall in relaxed standing position should be less than 5 cm.Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week
Global Perceived Effect Questionnaire: | six week
  Perceived effect of the intervention will be assessed by using the Global Perceived Effect Questionnaire (GPE), a 5-point Likert-type scale evaluating the subjective self-reported improvement or deterioration after the intervention. GPE is widely used in the physical therapy literature. Assessment to be done at baseline, after 1st session, at 3rd week and at 6th week

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Islamabad Physiotherapy and Rehabilitation Centre (IPRC), Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No